CLINICAL TRIAL: NCT03433586
Title: COMT on Aspirin Platelets Effects (CAPE)
Acronym: CAPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kathryn Tayo Hall, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015D006250; K01HL130625 (NIH)
Record Dates: First submitted 2018-02-09; First posted 2018-02-14 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: participants will be randomized to aspirin or placebo
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pills that are visually identical to the Aspirin pills will be taken orally, daily for 10-14 days
  Interventions: Drug: Placebo
- Aspirin (Active Comparator): Aspirin (81mg) will be taken orally daily for 10-14 days.
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — 81mg of aspirin to be taken daily for 10-14 days
  Other Names: acetylsalicylic acid
  Arms: Aspirin
Drug: Placebo — Placebo pill (visually identical to aspirin pill) to be taken daily for 10-14 days
  Arms: Placebo

SUMMARY:
Specific Aim I: Examine the role of genetic variation in COMT on platelet function in a blinded, randomized, placebo controlled clinical trial of daily placebo or Aspirin (81mg) for 10 ± 3 days. Platelet function will be assessed with platelet aggregometry and by fluorescence-activated cell sorting (FACS) of platelet adhesion molecules P-selectin and GPIIb/IIIa in platelets activated with arachidonic acid, thrombin, collagen, epinephrine and ADP.

Specific Aim II: Examine the effects of platelet releasates harvested at the end of each treatment arm on angiogenesis.

DETAILED DESCRIPTION:
This is a randomized double-blinded, placebo controlled study. This study is designed to detect the variation in platelet function based on COMT variation and how these platelets respond to cancerous cells.

We expect to recruit 60 healthy participants with the intention of studying 45 participants to complete the protocol.

Individuals aged 18 to 40 years will be eligible to participate in this study if they do not have history of fainting/problems related to blood draws, major chronic medical illnesses, regular or current treatment of Aspirin™.

Examine the role of genetic variation in in catechol-O-methyltransferase (COMT) on platelet function in a randomized double-blinded placebo controlled clinical trial of daily Aspirin™ (81 mg) versus placebo over 10-14 days. Platelet function will be assessed with a platelet aggregometry and by fluorescence-activated cell sorting assessment of platelet adhesion molecule GPIIIb/IIIa and p-selectin.

ELIGIBILITY:
Inclusion Criteria:

* healthy, 18-40 years

Exclusion Criteria:

* taking aspirin. Smoking, pregnancy, history of cancer of cardiovascular disease. Mental illness.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
platelet aggregation | At end of treatment 10-14 days the platelets will be activated on the same day as blood collection.
  Platelets will be activated with arachidonic acid, thrombin, collagen, ADP and epinephrine

SECONDARY OUTCOMES:
% expression of P-selectin on resting and activated platelets | At end of treatment 10-14 days the platelets will be activated on the same day as blood collection.
  Platelets activated with arachidonic acid, ADP, collagen and epinephrine

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn T Hall, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The generation of large-scale human or non-human genome data is not an explicit plan in this proposal. However, any genomic data as it pertains to single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, or gene expression data produced from the work in this award will be made publicly available through the appropriate NIH data repositories including array express, Database of Genotypes and Phenotypes (dbGaP), Database of Short Genetic Variations (dbSNP) or Gene Expression Omnibus (GEO). We intend to share the results from this study in published manuscripts and presentations at National Meetings. Unique methodology or results developed or generated through this study will be made readily available for research purposes to qualified individuals within the scientific community. Interested researchers will be able to contact the corresponding authors of the publications for information about access to resources.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Hall KT, Nelson CP, Davis RB, Buring JE, Kirsch I, Mittleman MA, Loscalzo J, Samani NJ, Ridker PM, Kaptchuk TJ, Chasman DI. Polymorphisms in catechol-O-methyltransferase modify treatment effects of aspirin on risk of cardiovascular disease. Arterioscler Thromb Vasc Biol. 2014 Sep;34(9):2160-7. doi: 10.1161/ATVBAHA.114.303845. Epub 2014 Jul 17. PMID 25035343